CLINICAL TRIAL: NCT02434783
Title: The Relationship Between Peripheral Arterial Disease and Mitochondrial Respiratory Capacity
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/204
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Intermittent Claudication
Keywords: Blood circulation; Blood vessels; Mitochondria; Muscle, skeletal; Legs; Energy metabolism
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — gastrocnemicus muscle biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1st level of arterial insufficiency: asymptomatic PAD patients
- 2nd level of arterial insufficiency: Intermittent claudication patients
- 3rd level of arterial insufficiency: Critical limb ischemia patients
- No arterial insufficiency: Healthy individuals (control)

SUMMARY:
Current evidence cannot explain the clinical features of peripheral arterial disease only from the principle of reduced blood flow. Explanations have therefore in addition been linked to mitochondrial dysfunction of skeletal muscles.

This study will elucidate whether there is a relation between clinical variables of the different levels of arterial insufficiency in peripheral arterial disease and mitochondrial respiratory capacity.

ELIGIBILITY:
Inclusion Criteria:

* Asymptotic peripheral arterial disease (Ankle-brachial index < 0.9), intermittent claudication (Ankle-brachial index 0.4 - 0.9), or critical limb ischemia (Ankle-brachial index < 0.4)

Exclusion Criteria:

* Diagnosed with intermittent claudication secondary to vascular insufficiency
* Warfarin or heparin usage
* Underwent a vascular intervention in the last 6 months
* Active cancer, renal- or liver disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with arterial insufficience at 1 of three levels, either asymptotic, intermittent claudication or critical limb ischemia; and healthy persons in a control group
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
mitochondrial respiratory capacity | 1 hour
  measured in oxygen glux in pmol.s-1.mg-1, using mitochondrial respirometry on an Oxygraph-2k (Oroboros Instruments, Austria).

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Rognmo, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway